CLINICAL TRIAL: NCT06992037
Title: An Ambispective, Multicenter, Registry Study Comparing Clinical Outcomes of Participants Receiving Surgical Interventions for the Treatment of Nasal Airway Obstruction (The DUO Study)
Brief Title: An Ambispective Registry Study Comparing Clinical Outcomes of Surgical Interventions for the Treatment of Nasal Airway Obstruction.
Acronym: DUO
Status: Completed | Type: Observational
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP2144
Record Dates: First submitted 2025-04-09; First posted 2025-05-28 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Nasal Airway Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Functional Rhinoplasty: Patients received a non-study/Standard of Care Functional Rhinoplasty within the past 5 years
- Septoplasty: Patients received a non-study/Standard of Care Septoplasty within the past 5 years
- Vivaer: Patients received a Vivaer procedure (radiofrequency) within the past 5 years
- Rhinaer: Patients received a Rhinaer procedure (radiofrequency) within the past 5 years

SUMMARY:
The purpose of this study is to assess and compare the clinical outcomes associated with common surgical interventions for the treatment of nasal airway obstruction (NAO).

DETAILED DESCRIPTION:
This is a multicenter, ambispective registry study. The study will include assessment of prospective, long term outcomes by remote administration of patient reported outcome questionnaires. Participants identified in Part 1 of the study with outcomes available for at least 12 months following their surgical procedure for nasal airway obstruction will be identified by the treating physician and invited to participate in the long-term follow-up study. Participants agreeing to participate will be asked to complete a series of questions about their health experience following their surgery and will be asked to complete select health outcome questionnaires using a secure electronic survey platform.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 to 85 years old (inclusively).
* Sought treatment at the clinic for nasal airway obstruction.
* Had either a functional rhinoplasty or septoturbinoplasty within the time frame of January 01, 2013 to December 31, 2023 or a Temperature-Controlled Radiofrequency (TCRF) procedure between the dates of November 19, 2015 to December 31, 2023.
* Has access to a mobile device, tablet, or computer with internet access and has access to an email address.
* Willing and able to provide consent.
* Willing and able to complete the survey, including patient-reported outcome measures.
* Willing and able to comply with the patient-specific requirements outlined in the study protocol.

Exclusion Criteria:

* Had extreme nasal pathology or a history of extreme nasal injuries.
* Had cosmetic rhinoplasty with no functional component.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nasal airway obstruction that had either a functional rhinoplasty or septoturbinoplasty within the time frame of January 01, 2013 to December 31, 2023 or a TCRF procedure between the dates of November 19, 2015 to December 31, 2023.
Sampling Method: Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Scale (NOSE) Score | Jan 2013 - Dec 2025
  The NOSE survey is a disease-specific questionnaire designed to measure nasal obstruction. It is commonly used in otolaryngology practice to provide an objective measure of nasal obstruction. Patients rate on a 0-4 scale questions regarding congestion, ability to get air in nose during exercise, and others. Scores result in symptom severity classes of mild, moderate, severe or extreme NAO.
22-Item Sinonasal Nasal Outcome Test (SNOT-22) | Jan 2013 - Dec 2025
  The The Sino-Nasal Outcome Test (SNOT-22) Questionnaire is a validated patient-reported outcome measure established to delineate the presence and severity of sinonasal disorders. It is a widely used questionnaire for assessing the impact of chronic rhinosinusitis on a patient's quality of life.
  Minimum possible score: 0; Maximum possible score: 110. Higher scores indicate: A worse outcome, meaning more severe symptoms and a greater negative impact on quality of life.
Standard Cosmesis and Health Outcomes Survey (SCHNOS) | Jan 2013 - Dec 2025
  The SCHNOS survey is a validated 10-item survey with two-domains (nasal obstruction and nasal cosmesis) patient-reported outcomes survey designed to evaluate both functional and cosmetic components of rhinoplasty. Minimum possible score: 0, Maximum possible score: 40. Higher scores indicate: A better outcome, meaning improved nasal function and cosmesis.
Short Form-12 (SF-12 version 1) | Jan 2013 - Dec 2025
  SF-12 is a 12 question self-reported outcome measure assessing the impact of health on an individual's everyday life. It includes questions in 8 domains: limitations in physical activities due to health problems, limitations in social activities because of physical or emotional problems, limitations on usual role activities because of physical or emotional health problems, bodily pain, general mental health, vitality, and general health perceptions. A score above 50 indicates better than average health-related quality of life and scores less than 50 suggest below-average health. Minimum possible score: 0, Maximum possible score: 100. Higher scores indicate: A better outcome, meaning improved health-related quality of life
Mini-Rhinoconjunctivitis Quality of Life Score (Mini-RQLQ) | Jan 2013- Dec 2025
  The mini-RQLQ is a self-administered questionnaire that measures functional impairments that are most troublesome to adult patients because of their rhinoconjunctivitis. This instrument has 14 questions in 5 domains: activity limitation, practical problems, nose symptoms, eye symptoms and non-nose/eye symptoms). Minimum possible score: 0, Maximum possible score: 42. Higher scores indicate: A worse outcome, meaning more severe symptoms and a greater negative impact on quality of life.
Epworth Sleepiness Scale (ESS) | Jan 2013 - Dec 2025
  The ESS is a validated widely used self-administered screening questionnaire that evaluates excessive daytime sleepiness.
Change in Medication Dose | Jan 2013 - Dec 2025
  Change in the dose from prior to procedure to post procedure of medication used for treating Nasal Airway Obstruction Symptoms
Change in Medication Frequency | Jan 2013 - Dec 2025
  Change in the frequency of use (prior to procedure to post procedure) of medication used for treating Nasal Airway Obstruction Symptoms
Change in use of Nasal Airway Obstruction Devices | Jan 2013 - Dec 2025
  Change in use of devices used for Nasal Airway Obstruction from prior to procedure to Post Procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Chicago Nasal & Sinus Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided